CLINICAL TRIAL: NCT06161844
Title: A Phase 3, Randomized, Open-label, Parallel-group, Multicenter, Controlled Study to Evaluate Efficacy and Safety of Semaglutide Injection (HD1916) vs. Ozempic® as add-on to Metformin in Patients With Type 2 Diabetics Mellitus
Brief Title: Efficacy and Safety of Semaglutide Injection (HD1916) in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD1916-002
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide injection (HD1916) (Experimental): Up to 1.0 mg semaglutide (HD1916) Metformin ≥ 1500 mg/day
  Interventions: Drug: semaglutide injection (HD1916)
- Ozempic® (Active Comparator): Up to 1.0 mg semaglutide (Ozempic®) Metformin ≥ 1500 mg/day
  Interventions: Drug: Ozempic®

INTERVENTIONS:
Drug: semaglutide injection (HD1916) — Up to 1.0 mg semaglutide injected subcutaneously once-weekly for 32 weeks Other Name: HD1916
  Arms: Semaglutide injection (HD1916)
Drug: Ozempic® — Up to 1.0 mg semaglutide injected subcutaneously once-weekly for 32 weeks Other Name: Ozempic Injectable Product
  Arms: Ozempic®

SUMMARY:
To evaluate the similarity of the efficacy and safety of semaglutide injection (HD1916) vs. Ozempic® in patients with type 2 diabetes mellitus (T2DM) with poor blood glucose control after metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤75 years old;
2. Patients diagnosed with type 2 diabetes;
3. A stable dose of metformin hydrochloride is administered on the basis of diet and exercise before screening (the minimum dose of metformin hydrochloride should meet the following requirements: metformin hydrochloride dose ≥1500 mg/ day), the treatment lasted for ≥8 weeks;
4. At the time of screening, HbA1c ≥ 7.5% and ≤ 11.0% (local lab); At baseline, HbA1c ≥ 7.0% and ≤10.5% (central lab);
5. At the time of screening, BMI≥18.5 kg/m^2 and ≤35 kg/m^2;
6. The patient of potential fertility is willing and must use a reliable contraceptive method to avoid pregnancy of the female patient or the male patient's partner during the whole study period and for at least 3 months after the last dose;
7. The patient is able to understand the informed consent form, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Patients with type 1 diabetes or other special types of diabetes;
2. Treatment with any glucose-lowering agent other than metformin hydrochloride within 8 weeks before screening or during the screening/run-in period (≤7 total days allowed in the 8 weeks before screening) or use of GLP-1 or a dual - or multi-target agent containing GLP-1 within the past 3 months;
3. Patients who meet the contraindications of GLP-1 RA drugs and metformin hydrochloride drugs;
4. Known allergy to the investigational drugs or excipients;
5. Acute metabolic complications within 6 months before screening, including but not limited to: diabetic ketoacidosis (DKA), hyperglycemic hyperosmolar state (HHS), or lactic acidosis;
6. Have serious chronic diabetic complications, including but not limited to: proliferative diabetic retinopathy, severe nonproliferative diabetic retinopathy, suspected or confirmed history of macular edema, history of renal dialysis or renal transplantation, severe peripheral vascular disease (such as amputation, chronic foot ulcers, intermittent claudication, etc.), or significant autonomic neuropathy (such as urinary retention, orthostatic hypotension, diabetic diarrhea, etc.);
7. A history of two or more episodes of grade 3 hypoglycemia within 6 months before screening or grade 3 hypoglycemia (grade 3: a severe hypoglycemic event that requires assistance from another person for treatment, with altered consciousness, physical appearance, but without a specific glycemic cutoff) before screening to randomization;
8. Stress conditions such as severe trauma, acute infection or major surgery under general anesthesia that may affect blood glucose levels within 1 month before screening or during screening/induction;
9. Patients with hyperthyroidism or hypothyroidism at screening (except those with stable drug dose control for more than 3 months and normal thyroid function tests) or clinically significant abnormal thyroid function test results at screening and requiring drug treatment;
10. Patients with obvious blood system diseases that may cause hemolysis or red blood cell instability and affect HbA1c detection, including but not limited to: hemolytic anemia, aplastic anemia, myelodysplastic syndrome, etc., or blood donation or blood loss ≥400 mL within 4 weeks before screening, or receiving blood transfusion;
11. Have undergone metabolic surgery prior to screening, or had used medications and/or supplements with approved weight-loss indications within 3 months;
12. Patients with severe heart disease or cardiac insufficiency. Including, but not limited to, decompensated heart failure (NYHA class Ш or Ⅳ); Uncontrolled or severe arrhythmia; Patients have a history of acute myocardial infarction, unstable angina pectoris, or coronary stent implantation, coronary artery bypass grafting, or coronary angioplasty within 6 months before screening;
13. Patients with incident cerebrovascular events (including, but not limited to, ischemic stroke, hemorrhagic stroke, and transient ischemic attack) within 6 months prior to screening;
14. Uncontrolled hypertension (defined as systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg), or hypotension (blood pressure < 90/60mmHg at screening);
15. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2) at screening;
16. Patients with a history of severe chronic gastrointestinal disease, clinically significant abnormal gastric emptying (e.g., diabetic gastroparesis, pyloric stenosis, etc.), long-term use of drugs that directly reduce gastrointestinal peristalsis, or those who have undergone gastrointestinal resection;
17. Patients with a history of chronic pancreatitis or idiopathic acute pancreatitis, or with obvious signs and symptoms of pancreatitis at the time of screening, or who have undergone pancreatectomy;
18. Treatment with systemic glucocorticoids (other than inhaled or topical glucocorticoids) within 4 weeks before screening;
19. Laboratory values at screening or before randomization:

    1. fasting blood glucose ≥13.9mmol/l;
    2. ALT and/or AST > 3× upper limit of normal (ULN);
    3. serum calcitonin >ULN;
    4. estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m^2 (estimated using CKD-EPI formula);
    5. hemoglobin (Hgb) <100 g/L;
    6. fasting triglyceride (TG) ≥5.7mmol/L;
    7. serum amylase and/or lipase > 3×ULN (if lipase cannot be detected in some centers, it is acceptable to judge based on amylase only);
20. Prolonged QTc interval (QTc interval >450 msec in men and >460 msec in women) on 12-lead electrocardiogram at screening or before randomization; PR interval >220 ms; (QTc values need to be corrected by QTcF formula);
21. Serologic examination:

    1. human immunodeficiency virus antibody or treponema pallidum antibody positive;
    2. hepatitis C antibody positive;
    3. hepatitis B surface antigen (HBsAg) is positive, and the quantitative test result of hepatitis B virus DNA is higher than the upper limit of the reference range;
22. Patients with a history of drug abuse, drug use, or alcohol dependence;
23. History of malignant tumor;
24. Women who are pregnant, lactating or have a positive pregnancy test;
25. Patients who participated in other clinical trials within 3 months before screening and received the last study medication within 3 months;
26. Patients who had other factors, as judged by the investigator, that precluded participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 32 in glycosylated haemoglobin (HbA1c) | Week 32

SECONDARY OUTCOMES:
Change from baseline to week 20 in HbA1c | Week 20
Change from baseline to week 20, 32 in fasting blood glucose | Week 20 and 32
Percentage of participants who achieved HbA1c < 7.0% and HbA1c ≤6.5% at week 20 or week 32 | Week 20 and 32
Change from baseline to week 20, 32 in body weight | Week 20 and 32
Change from baseline to week 20, 32 in postprandial blood glucose | Week 20 and 32
Percentage of participants who were offered rescue medication at week 20 | Week 32
Incidence and severity of adverse events | Week 35
Occurence of anti-semaglutide antibodies and neutralizing antibody | Week 35
Blood concentration of semaglutide | Week 35

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No